CLINICAL TRIAL: NCT00207935
Title: Use of Sustained Release Antiepileptic Medication (Depakote® ER) for Pediatric Epilepsy in a Mental Retardation/Developmental Disorder Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNMC IRB 3579
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2008-05-05 (Estimated); Status verified 2005-09

CONDITIONS: Epilepsy; Mental Retardation; Developmental Disabilities
Keywords: Seizures; Depakote; Developmental Delay; Mental Retardation; Swallow
MeSH Terms: conditions — Epilepsy; Intellectual Disability; Developmental Disabilities; Seizures; Learning Disabilities

INTERVENTIONS:
Behavioral: Swallow instruction

SUMMARY:
This study is being done to see if children with learning problems can learn how to swallow pills without chewing them. The reason this is important is that if a person has seizures, medications must be taken every day. Most medications need to be taken 2 or 3 times per day. Some medications have slow release and only are taaken once per day. Medications with slow release usually come in capsule form and cannot be opened or chewed. This study investiates whether children with developmental delay can be taught how to swalow pills.

DETAILED DESCRIPTION:
Participants will initially be consented into the study, and receive baseline assessments. At the baseline visit, seizure types (partial, primary generalized, secondary generalized), seizure foci localization, and additional medication treatment status for the duration of the study will be established. IQ status which has been done (either by the school system or as part of a developmental assessment,) will be used.

Behavioral status will be verified and related to seizure activity as well. Behavioral measures will include the Vineland (a measure of life skills assessment) and the Child Behavior Checklist. Participants then return for a study visit two weeks later. At that time initial laboratory tests will be done including a trough level of valproic acid. Pregnancy tests will be done on all females of childbearing potential, because of the known risk of valproic acid during pregnancy. Participants will return for a third study visit two weeks later where another trough valproic acid level will be obtained, and effective dosage conversion of Depakote® Sprinkle to Depakote® ER will occur. Subsequent study visits will occur at weeks 6 and 8 (2 and 4 weeks respectively, after the dose conversion); trough valproic acid levels will be obtained each time. At each study visit, neurologic (seizure control) and behavioral status will be reviewed as well as monitoring for side effects and adverse events. Each study visit will also include instruction and coaching regarding strategies for pill swallowing and other aspects of adherence to treatment regimen. Compliance will be ascertained by means of drug level monitoring pre and post dosage conversion. Clinical global improvement in functioning for both behavioral issues and epilepsy will be assessed.

The study will conclude after the 5th visit.

Table of Events Visit 1 2 3 4 5 Day -28 -14 0 14 28 Week -4 -2 0 2 4 Informed Consent X Eligibility Criteria X X Demographics X Medical and Surgical History X IQ verification X QOLIE X X Vineland X X CBCL X X Seizure assessment X X X X X Physical and Neurologic exam X X X VS X X X Lab assessments X X

ELIGIBILITY:
Inclusion Criteria:

1. Age 4-18 years, inclusive.
2. Clinical Diagnosis of Partial or Primary Generalized Seizure Disorder
3. Documented IQ scores in the range of borderline, mild, moderate, or severe mental retardation (IQ<80).
4. Currently Treatment regimen includes Depakote® Sprinkles either as monotherapy or adjunctive therapy. Dosages should have been stable for at least 4 weeks prior to baseline.
5. Subject's parent or guardian must be capable of maintaining a record of dosing times, seizure characteristics, and adverse events.

Exclusion Criteria:

1. Oral Motor Dysfunction to the degree that swallowing is affected.
2. History of significant aspiration.
3. Serious medical conditions such as cancer, pancreatitis, diabetes, HIV.
4. History of hepatic dysfunction including history of elevated liver enzymes (AST or ALT values greater or equal to three times the upper limit of normal).
5. History of metabolic disorders including urea cycle disorders.
6. Pregnancy

   -

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-08; Study Completion 2007-03

PRIMARY OUTCOMES:
Ability to swallow capsules in a mentally retarted developmentally delayed population

CONTACTS AND LOCATIONS:
Overall Officials: Joan A Conry, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States